CLINICAL TRIAL: NCT00078286
Title: Safety and Efficacy of Sertraline for Depression CHF
Brief Title: Antidepressant Medication Treatment for Depression in Individuals With Chronic Heart Failure
Acronym: SADHART-CHF
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00010340; R01MH063211 (NIH); DATR A4-GPX
Record Dates: First submitted 2004-02-20; First posted 2004-02-24 (Estimated); Results first posted 2013-02-27 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-01

CONDITIONS: Heart Failure, Congestive; Chronic Heart Failure; Depression
Keywords: Antidepressive Agents
MeSH Terms: conditions — Heart Failure; Depression | interventions — Sertraline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sertraline (Experimental): Participants will take sertraline for 12 weeks
  Interventions: Drug: Sertraline
- Placebo (Placebo Comparator): Participants will take placebo for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sertraline — Dosage ranging from 50 mg to 200 mg once a day
  Other Names: Zoloft
  Arms: Sertraline
Drug: Placebo — Dosage ranging from 50 mg to 200 mg once a day
  Other Names: Inactive pill
  Arms: Placebo

SUMMARY:
This study will examine the effect of antidepressant medication on rates of death and disease in depressed people with chronic heart failure.

DETAILED DESCRIPTION:
Comorbid depression in people with chronic medical illness is a serious public health concern. Depressive disorders lead to increased morbidity, mortality, and poorer outcomes in ischemic heart disease, a leading cause of chronic heart failure (CHF). Evidence suggests that a relationship exists between depression and CHF; studies that examine the way CHF is affected by depression treatments are needed.

Participants in this study will be randomly assigned to receive either sertraline or placebo for 12 weeks. Assessments will be made at Weeks 2, 4, 6, 8, 10, and 12. Participants who do not respond to their treatment will have their medication dose adjusted following assessment. Interviews and rating scales will be used to assess depressive symptoms, cognitive status, psychiatric comorbidity, daily and chronic stress, and social support. A follow-up visit will take place 6 months, 1 year, 2 years, and 3 years after study completion.

ELIGIBILITY:
Inclusion Criteria:

* Chronic heart failure
* Diagnostic and Statistical Manual- Fourth Edition (DSM-IV) criteria for major depression
* Current use of any antipsychotic medication at study entry

Exclusion Criteria:

* Life-threatening comorbidity with a 50% or higher likelihood of death within 1 year
* History of psychoses, bipolar disorder, or severe personality disorder
* History of alcohol or drug dependence in the last year
* Severe physical disability that may interfere with the study
* Neurological impairment
* Active suicidal ideations
* Current use of antidepressant medication(s) at the start of study medication

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 469 (Actual)
Dates: Start 2003-11; Primary Completion 2008-03 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ranga Krishnan, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Result] O'Connor CM, Jiang W, Kuchibhatla M, Silva SG, Cuffe MS, Callwood DD, Zakhary B, Stough WG, Arias RM, Rivelli SK, Krishnan R; SADHART-CHF Investigators. Safety and efficacy of sertraline for depression in patients with heart failure: results of the SADHART-CHF (Sertraline Against Depression and Heart Disease in Chronic Heart Failure) trial. J Am Coll Cardiol. 2010 Aug 24;56(9):692-9. doi: 10.1016/j.jacc.2010.03.068. PMID 20723799
- [Derived] Xiong GL, Prybol K, Boyle SH, Hall R, Streilein RD, Steffens DC, Krishnan R, Rogers JG, O'Connor CM, Jiang W; SADHART-CHF Investigators. Inflammation Markers and Major Depressive Disorder in Patients With Chronic Heart Failure: Results From the Sertraline Against Depression and Heart Disease in Chronic Heart Failure Study. Psychosom Med. 2015 Sep;77(7):808-15. doi: 10.1097/PSY.0000000000000216. PMID 26186432
- [Derived] Steffens DC, Wei Jiang, Krishnan KR, Karoly ED, Mitchell MW, O'Connor CM, Kaddurah-Daouk R. Metabolomic differences in heart failure patients with and without major depression. J Geriatr Psychiatry Neurol. 2010 Jun;23(2):138-46. doi: 10.1177/0891988709358592. Epub 2010 Jan 25. PMID 20101071
- [Derived] Jiang W, O'Connor C, Silva SG, Kuchibhatla M, Cuffe MS, Callwood DD, Zakhary B, Henke E, Arias RM, Krishnan R; SADHART-CHF Investigators. Safety and efficacy of sertraline for depression in patients with CHF (SADHART-CHF): a randomized, double-blind, placebo-controlled trial of sertraline for major depression with congestive heart failure. Am Heart J. 2008 Sep;156(3):437-44. doi: 10.1016/j.ahj.2008.05.003. Epub 2008 Jul 7. PMID 18760123

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in November, 2003 and concluded in March, 2008. Subjects were recruited from cardiology inpatient units as well as outpatient cardiology clinics.
Period: Overall Study
Arm/Group | Sertraline | Placebo
Started | 234 | 235
Completed | 138 | 152
Not Completed | 96 | 83

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sertraline | Placebo | Total
Number analyzed (Participants) | 234 | 235 | 469
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0.0
  Between 18 and 65 years | 131 | 147 | 278.0
  >=65 years | 103 | 88 | 191.0
Age Continuous [Mean (Standard Deviation); unit: years] | 62.9 (10.5) | 61.4 (11.1) | 62.1 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 89 | 190.0
  Male | 133 | 146 | 279.0

OUTCOME MEASURES:

1. Primary Outcome: Symptoms of Depression in Congestive Heart Failure Patients With Clinical Depression After Treatment With Sertraline or Placebo
Description: Symptoms of depression (as measured by the Hamilton Depression Rating Scale, HDRS) in congestive heart failure patients with clinical depression after treatment with sertraline or placebo.
  The 17-item Hamilton Depression Rating Scale (HDRS) is a rater-administered assessment of depression severity, with total score ranges from 0 (not at all depressed) to 52 (most severely depressed). Change in depression was measured as the difference between the 12-week HDRS scores and the baseline HDRS scores. Thus, a negative value reflects an improvement in depressive symptoms over the 12-week period.
Time Frame: Measured at Week 12
Population: Analysis was based on intent to treat (ITT), using random coefficient modeling.
Measure: Mean (Standard Deviation); unit: HDRS Change Score
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 234 | 235
HDRS Change Score | -7.1 (0.5) | -6.8 (0.5)
Statistical Analysis 1: Comparison: Sertraline vs Placebo; A hierarchical mixed model was used, analyzing the fixed effects of treatment, the natural log of time, natural log of time squared, the interactions of time and time squared with treatment and site, as well as the random effects of patient, patient-by-time, and square of patient-by-time; Test type: Non-Inferiority or Equivalence — *Power analysis already provided; p = 0.89, Mixed Models Analysis; Significance was tested at p=.05; Difference in mean change score = -0.3

2. Secondary Outcome: Percentage of Cardiac Events and Morbidity / Mortality, Including Rehospitalization, in Congestive Heart Failure Patients With Depression After Treatment With Sertraline or Placebo.
Description: Composite cardiovascular scores are calculated for each participant using recorded cardiac events, morbidity/mortality, rehospitalization, and discontinuation due to cardiovascular events. Composite score is compared for sertraline and placebo treatment groups.
Time Frame: Measured at Week 12
Population: Analysis was based on intent to treat (ITT).
Measure: Number; unit: percentage of participants
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 138 | 152
percentage of participants
  Cardiovascular Status Worsened | 29.9 | 31.1
  Cardiovascular Status Improved | 40.6 | 43.8
  Cardiovascular Status Unchanged | 29.5 | 25.1
Statistical Analysis 1: Comparison: Sertraline vs Placebo; Tests for differences of proportions were used to examine the composite cardiovascular status outcome at the end of acute treatment. Chi-square tests were used to test for overall treatment differences, with a Mantel Haenszel test performed to examine treatment differences when controlling for clinical site. The primary analyses were conducted on the tri-level cardiovascular status outcome; Test type: Superiority or Other; p = .78, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.08

ADVERSE EVENTS:
Time Frame: 12-weeks
Description: All participants were followed via phone or mail to ascertain clinical events and vital status every 2 weeks during the 12-week treatment phase. The national death index was used to ascertain vital status of participants who could not be reached via phone or mail.
Groups:
- Sertraline: Serious adverse events in Sertraline Arm
- Placebo: Serious adverse events in Placebo Arm
Arm/Group | Sertraline | Placebo
Serious Adverse Events (participants affected / at risk) | 57/234 | 63/235
Other Adverse Events (participants affected / at risk) | 22/234 | 23/235
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sertraline (N=234) | Placebo (N=235)
Cardiovascular (Cardiac disorders) | 40 (69) | 44 (72)
Psychiatric (Psychiatric disorders) | 0 (0) | 2 (2)
Noncardiovascular and nonpsychiatric (General disorders) | 17 (29) | 17 (22)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.80% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sertraline (N=234) | Placebo (N=235)
Congestive Heart Failure (Cardiac disorders) | 11 (19) | 10 (20)
Unstable Angina (Cardiac disorders) | 2 (5) | 2 (5)
Other Cardiovascular (Cardiac disorders) | 9 (12) | 11 (16)

LIMITATIONS AND CAVEATS:
NFS may have limited our ability to detect effect of sertraline on depression scores. Dropout rate was higher than expected. A 12-week duration of therapy may have been insufficient to show potential effects of sertraline on clinical outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No